CLINICAL TRIAL: NCT04930796
Title: Randomized Open-label Study to Evaluate the Pharmacokinetics and Safety of VER-01 After Single Dose With and Without Meal in Healthy Volunteers
Brief Title: Food Effect Study of VER-01 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VER-PK-002
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: THC; Tetrahydrocannabinol; Cannabis; Pharmacokinetics
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VER-01 following overnight fast (Day 1) and a high-fat breakfast (Day 4) (Experimental): The PK profile of VER-01 is investigated after oral intake of a single dose VER-01 (corresponding to 10 mg THC) in the morning after a 10-hour fasting period on day 1, and 30 minutes after the intake of a standardised high-fat breakfast has been started on day 4 (Group 1).
  Interventions: Drug: VER-01
- VER-01 following a high-fat breakfast (Day 1) and overnight fast (Day 4) (Experimental): The PK profile of VER-01 is investigated after oral intake of a single dose VER-01 (corresponding to 10 mg THC) in the morning 30 minutes after the intake of a standardised high-fat breakfast has been started on day 1 and after a 10-hour fasting period on day 4 (Group 2).
  Interventions: Drug: VER-01

INTERVENTIONS:
Drug: VER-01 — standardised cannabis extract (containing 21 mg THC per gram drug product)

SUMMARY:
Evaluation of pharmacokinetics, tolerability and safety of VER-01 depending on the intake a high-fat meal in healthy volunteers

DETAILED DESCRIPTION:
Determination of the effect of food intake on the pharmacokinetic (PK) profile of VER-01 in healthy volunteers.

Group 1: 9 subjects receive VER-01 (corresponding to 10 mg THC) in the morning after a 10-hour fasting period on day 1, and 30 minutes after the intake of a standardised high-fat breakfast has been started on day 4.

Group 2: 9 subjects receive VER-01 (corresponding to 10 mg THC) in the morning after 30 minutes after the intake of a standardised high-fat breakfast has been started on day 1 and after a 10-hour fasting period on day 4.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers
* Age: 18-45 years
* BMI: 19-30 kg/m²
* Body weight ≥ 50 kg
* volunteers in good general condition based on medical history, physical examination, resting ECG and clinical laboratory tests
* Willingness of men to use a reliable method of contraception and not to donate sperm during and at least 3 months after the last intake of the study product
* Understanding of the German language, ability to give consent and compliance
* The subject has understood the instructions to avoid changes in lifestyle and eating habits
* Signed patient information and consent form of the study participant
* Study participant can stick to the diet plan, especially high-fat breakfast

Exclusion Criteria:

* Consumption of cannabis-based products within 30 days prior to study start
* Well-known strong adverse events in connection with cannabis consumption
* Known allergy to cannabis, sesame seeds, or derivative products
* alcohol/drug/medication abuse or physical dependence on opioids, barbiturates, amphetamines, cocaine or benzodiazepines within the last 10 years or current intake of methadone
* Positive drug test for illegal substances and/or alcohol test at time T0
* Heavy smokers (>10 cigarettes/day)
* Heavy caffeine consumers (>450 mg caffeine/day equal to approx. 5-6 cups of filter coffee)
* Drastic change in diet within 30 days before study start
* Mental illness (psychoses, schizophrenia, bipolar disorder, severe depression, anxiety disorder, suicide)
* Mental illness (psychoses, schizophrenia, bipolar disorder, severe depression, anxiety disorder, suicide) in a first-degree relative (parents and children)
* subjects with orthostatic hypotension during screening (drop in systolic blood pressure by ≥20 mmHg after change of position)
* Cardiovascular event within the last 3 months, untreated hypertension, untreated hypothyroidism, surgery within the last 2 months
* cardiac insufficiency
* Subjects with a serious disease or disorder which, in the opinion of the investigator, does not allow safe participation in the study from a medical point of view
* Intake of prescription drugs within the last 14 days, OTC test products within the last 7 days before the start of the study or during the study period
* Eating of grapefruit products is not allowed during the study and 10 days before the first intake of the study product
* Participation in another clinical trial in the period of 90 days before the start of the trial
* Existing desire to have children or planned sperm donation (within the duration of the study and 3 months after end of the study)
* Planned blood donation
* No ability to consent
* Subject is in a dependency/employment relationship with the sponsor or investigator or other persons who may be under pressure.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - AUC 0-t | On Day 1 and Day 4
  Analysis of AUC 0-t (AUC from time 0 to 24 hours) of THC over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - AUC 0-∞ | On Day 1 and Day 4
  Analysis of AUC 0-∞ (AUC from time 0 extrapolated to infinity) of THC over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC] - C max | On Day 1 and Day 4
  Analysis of C max (maximum plasma concentration) of THC over a defined period of time in dependance of a high-fat meal.

SECONDARY OUTCOMES:
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - AUC 0-t | On Day 1 and Day 4
  Analysis of AUC 0-t (AUC from time 0 to 24 hours) of 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - AUC 0-∞ | On Day 1 and Day 4
  Analysis of AUC 0-∞ (AUC from time 0 extrapolated to infinity)of 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - C max | On Day 1 and Day 4
  Analysis of C max (maximum plasma concentration) of 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - λ z | On Day 1 and Day 4
  Analysis of λ z (terminal elimination constant) of THC, 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - t 1/2 | On Day 1 and Day 4
  Analysis of t 1/2 (elimination half-life) of THC, 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - T max | On Day 1 and Day 4
  Analysis of T max (time to reach Cmax)of THC, 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - C L/F | On Day 1 and Day 4
  Analysis of C L/F (plasma clearance) of THC, 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.
Pharmacokinetic profile of Δ9-tetrahydrocannabinol [THC], 11-Hydroxy-Δ9-tetrahydrocannabinol [11-OH-THC] and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol [THC-COOH] - V area/F | On Day 1 and Day 4
  Analysis of V area/F (volume of distribution) of THC, 11-OH-THC and THC-COOH over a defined period of time in dependance of a high-fat meal.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Professor, Principal Investigator — University of Medicine in Vienna - Department of Clinical Pharmacology
Locations (1):
- University of Medicine in Vienna - Department of Clinical Pharmacology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No